CLINICAL TRIAL: NCT01897246
Title: Computer Assisted Planning of Corrective Osteotomy for Distal Radius Malunion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Collaborators: AO Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10.0363
Record Dates: First submitted 2012-06-11; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Extra-articular Distal Radius Malunions
Keywords: distal radius malunion; extra-articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-assisted pre-operative planning (Active Comparator): Patients enrolled in this arm will undergo corrective surgery of the distal radius, with pre-operative computer-assisted planning and virtual osteotomy.
  Interventions: Procedure: Corrective osteotomy with computer-assisted pre-operative planning
- Conventional pre-operative planning (Active Comparator): Patients in this group will undergo corrective osteotomy of the distal radius wit conventional pre-operative planning.
  Interventions: Procedure: Corrective osteotomy with conventional preoperative planning

INTERVENTIONS:
Procedure: Corrective osteotomy with computer-assisted pre-operative planning — The corrective osteotomy will be planned with computer-assisted pre-operative planning and virtual osteotomy.
  Arms: Computer-assisted pre-operative planning
Procedure: Corrective osteotomy with conventional preoperative planning — The corrective osteotomy will be planned with conventional preoperative planning.
  Arms: Conventional pre-operative planning

SUMMARY:
The investigators are comparing post-operative patient-rated functional outcome between patients who undergo corrective osteotomy for extra-articular malunited distal radius fractures with and without computer assisted pre-operative planning and virtual osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 18 yrs of age)
* Extra-articular malunion of the distal radius
* Fluent in English

Exclusion Criteria:

* Pregnant patients
* prisoners
* patients with impaired decision making ability
* patients with a bony deformity in the distal forearm contralateral to the one with distal radius malunion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Grip Strength | Up to 12 months
  Grip strength as compared to the normal, contralateral hand is considered the most important outcome measure for patients with distal radius fractures.

SECONDARY OUTCOMES:
Range of motion | Up to 12 months
DASH Questionnaire | Up to 12 months
Mayo Wrist score | Up to 12 months
Gartland and Werley score | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rodrgio Moreno, MD, Principal Investigator — Christine M. Kleinert Institute of Hand and Microsurgery
Locations (1):
- Christine M. Kleinert Institute of Hand and Microsurgery, Louisville, Kentucky, United States